CLINICAL TRIAL: NCT01041521
Title: The Impact of Omega Three Fatty Acids on Vascular Function in HIV
Acronym: HOST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVZ112667; 1R01HL096585-01A1 (NIH)
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: High Triglyceride Level; HIV Infection
Keywords: HIV infection; Dyslipidemia; Elevated Triglyceride level; vascular function (BART); arterial stiffness; omega three fatty acids; complementary therapies
MeSH Terms: conditions — HIV Infections; Dyslipidemias | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovaza (omega three fatty acid) (Experimental): Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks.
  Other Names:
  Lovaza was previously known as Omacor (omega-3-acid ethyl esters) capsules
  Interventions: Drug: Lovaza
- sugar pill (No Intervention): Dietary Supplement: sugar pill
  2 capsules given twice daily Arms: sugar pill

INTERVENTIONS:
Drug: Lovaza — Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 24 months
  Other Names: omega three fatty acids; previously known as Omacor
  Arms: Lovaza (omega three fatty acid)

SUMMARY:
The study seeks to determine if the use of omega three fatty acids in individuals infected with HIV and with high triglycerides leads to improved triglyceride levels, better blood vessel function and decrease in the amount of obstruction in blood vessels.

DETAILED DESCRIPTION:
While omega-three fatty acids have been shown to be beneficial for triglycerides (TG) and HDL-C levels in HIV uninfected individuals and in some small, short duration studies in HIV-infected individuals, there are no data that extend these observations to determine whether intake of omega-three fats over a more prolonged time period will also have a beneficial impact on functional outcomes such as vascular endothelial function and anatomic surrogate markers of cardiovascular disease (CVD) in HIV-infected patients.

We propose a randomized, double blind trial of purified omega-three fatty acids in HIV-infected individuals with elevated levels of triglycerides. While the impact of omega-three fatty acids on lipid profiles should be evident early (within 12 weeks); we propose to conduct this trial for a full 24 months to test our overall hypothesis that this intervention will not only improve triglyceride and HDL-C levels, improve HDL-subpopulations, plasma and membrane phospholipids and decrease inflammation, but will also improve brachial artery reactivity testing (BART) as a measure of vascular endothelial function at 24 weeks and 24 months and arterial stiffness measured by a pulse wave velocity test as a surrogate marker of CVD risk at 24 months when compared to controls.

The specific aims of this proposal include:

1. To conduct a randomized, placebo controlled trial of omega-three fatty acids over 24 months in HIV-infected individuals with elevated levels of triglycerides (> 150 mg/dl).
2. To demonstrate the impact of omega-three fatty acid intake on TG levels and on HDL-C levels, HDL subpopulations, composition of plasma and membrane phospholipids, and chronic inflammation as measured by c-reactive protein (CRP), sPLA2 and by levels of arachidonic acid.
3. To demonstrate the impact of omega-three fatty acid intake on BART at 24 weeks and 24 months and on arterial stiffness at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected men and women at least 18 years of age,
* On stable HAART for the previous two months and without anticipated changes in their HAART regimen throughout the duration of the study,
* Fasting triglycerides > 150 mg/dl and < 2,500 mg/dl
* Participants may be on lipid lowering therapy; if on lipid lowering therapy, therapy must be stable for 8 weeks and cannot be changed during the course of the study.
* Participants may be on beta blockers (e.g., Atenolol, Metoprolol, Propranolol), and Estrogens (e.g., Estinyl; Estrace; Estraderm), however therapy with these agents must be stable for 8 weeks before starting the study and cannot be altered while on study unless deemed medically necessary by the participant's medical provider and approved by Dr. Wanke.
* Female participants of reproductive age must not be pregnant (negative test) or lactating at screening and throughout the trial and agree to use contraception for the course of the trial and 2 months after the trial unless they are surgically sterilized (tubal ligation or hysterectomy), or post-menopausal with no menses for > 1 year.
* Ability to provide consent.

Exclusion Criteria:

* plasma HIV-1 RNA > 10,000 copies/ml
* change in HAART regimen over two months prior to study entry
* change in lipid lowering therapy within 2 months (8 weeks)
* Pregnancy in female participants
* Evidence of liver or renal disease with values of liver enzymes > 5 X upper limit of normal or creatinine > 1.5 X upper limit of normal
* presence of active opportunistic infection or malignancy
* presence of other inflammatory or end organ disease (, rheumatoid arthritis, active treatment for hepatitis c, or other diseases that may alter inflammatory markers)
* routine ingestion of fish oil (individuals who have used fish oil would be reconsidered for study participation if they discontinue use of fish oil for 8 weeks and TG levels remain elevated).
* Allergic to fish or Lovaza
* BMI >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-01; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Wanke, MD, Principal Investigator — Tufts University
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants were enrolled but the did not participate due to 1) declining to participate, 2) inability of study team to locate participant, or 3) moving out of state.
Groups:
- Lovaza (Omega Three Fatty Acid): Lovaza: Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 24 months
  Other Names:
  Lovaza was previously known as Omacor (omega-3-acid ethyl esters) capsules
- Sugar Pill: Dietary Supplement: sugar pill
  2 capsules given twice daily for 24 months
Period: Overall Study
Arm/Group | Lovaza (Omega Three Fatty Acid) | Sugar Pill
Started | 61 | 56
Completed | 44 | 40
Not Completed | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Lovaza (Omega Three Fatty Acid): Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks.
  Other Names:
  Lovaza was previously known as Omacor (omega-3-acid ethyl esters) capsules
  Lovaza: Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 24 months
- Total: Total of all reporting groups
Arm/Group | Lovaza (Omega Three Fatty Acid) | Sugar Pill | Total
Number analyzed (Participants) | 61 | 56 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9) | 50 (9) | 51 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 46 | 46 | 92
Region of Enrollment [Number; unit: participants]
  United States | 61 | 56 | 117
Current smoker [Count of Participants; unit: Participants] | 24 | 16 | 40
CD4+ cell count [Mean (Standard Deviation); unit: cells/cubic mL] | 652 (394) | 644 (309) | 648 (354)
Undetectable HIV viral load [Count of Participants; unit: Participants] | 58 | 52 | 110
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/meters squared] | 28 (6) | 28 (6) | 28 (6)

OUTCOME MEASURES:

1. Primary Outcome: Triglyceride Level
Time Frame: 24 months
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Lovaza (Omega Three Fatty Acid) | Sugar Pill
Number analyzed (Participants) | 43 | 40
mg/dL | 130 [100 to 166] | 159 [118 to 233]

2. Secondary Outcome: Vascular Function
Description: Carotid-femoral pulse wave velocity is a measure of arterial stiffness, with lower values indicating less arterial stiffness.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Lovaza (Omega Three Fatty Acid) | Sugar Pill
Number analyzed (Participants) | 41 | 40
m/s | 833 (238) | 832 (152)

ADVERSE EVENTS:
Arm/Group | Lovaza (Omega Three Fatty Acid) | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 22/61 | 21/56
Other Adverse Events (participants affected / at risk) | 27/61 | 16/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza (Omega Three Fatty Acid) (N=61) | Sugar Pill (N=56)
excessive burping/gas, reflux (Gastrointestinal disorders) | 2 (3) | 0 (0)
nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Leg swelling or edema (Vascular disorders) | 0 (0) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
sepsis (Infections and infestations) | 1 (2) | 0 (0)
Pleural fluid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — "fluid around lungs"
stroke (Nervous system disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
asthma/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
heart failure (Cardiac disorders) | 0 (0) | 3 (4)
myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
orthopedic surgery (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
death (Cardiac disorders) | 0 (0) | 1 (1) — MI and renal failure
chest pain (Cardiac disorders) | 0 (0) | 3 (3)
diabetic incident (Endocrine disorders) | 0 (0) | 2 (4)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
elevated triglycerides (General disorders) | 1 (1) | 1 (1)
Infection of urinary tract (Infections and infestations) | 2 (2) | 1 (1)
renal failure/elevated creatinine (Renal and urinary disorders) | 0 (0) | 2 (2)
joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
difficulty swallowing (Gastrointestinal disorders) | 0 (0) | 1 (1)
tension headache (Nervous system disorders) | 1 (1) | 0 (0)
numbness (Nervous system disorders) | 1 (1) | 1 (1)
sciatic nerve/muscle spasm (Nervous system disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
acute/chronic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
prostate resection due to prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
concussion (Nervous system disorders) | 1 (1) | 0 (0)
epiglottitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
confusion (Nervous system disorders) | 0 (0) | 1 (1)
cocaine-induced bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
False positive TB test (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
viral gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
broken denture (General disorders) | 0 (0) | 1 (1)
hernia repair (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever and cough (Infections and infestations) | 0 (0) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
liver infection (Infections and infestations) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
cardiac bypass surgery (Cardiac disorders) | 1 (1) | 0 (0)
foot infection (Infections and infestations) | 1 (1) | 0 (0)
rash/eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza (Omega Three Fatty Acid) (N=61) | Sugar Pill (N=56)
excessive gas / burping /bloating (Gastrointestinal disorders) | 9 (10) | 4 (4)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
body aches (General disorders) | 1 (1) | 0 (0)
Diarrhea or loose stools (Gastrointestinal disorders) | 8 (9) | 5 (5)
elevated total bilirubin (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
leg swelling and edema (Vascular disorders) | 3 (4) | 2 (2)
rash or hives (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
asthma/pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
total body itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
surgery (rectal/bladder, hernia) (General disorders) | 1 (1) | 1 (1)
body odor (General disorders) | 0 (0) | 1 (1)
change in taste (General disorders) | 1 (1) | 0 (0)
dehydration (General disorders) | 1 (1) | 0 (0)
pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — torso above breast
concussion (Nervous system disorders) | 0 (0) | 1 (1)
kidney stent (Renal and urinary disorders) | 1 (1) | 0 (0)
wrist sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
sacral fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
increased abdominal fat (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fall with loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
fever (General disorders) | 1 (1) | 0 (0)
fluid in ears (Ear and labyrinth disorders) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
PLEASE NOTE THAT THE PRINCIPLE INVESTIGATOR (CHRISTINE WANKE) HAS LEFT TUFTS UNIVERSITY IN RETIREMENT AND CANNOT BE CONTACTED. PLEASE ALSO NOTE THAT THIS IS NOT AN "APPLICABLE CLINICAL TRIAL". - 9/3/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No